CLINICAL TRIAL: NCT01546623
Title: A Phase 3, Multi-center, Randomized, Open-label, Parallel-group, Comparative Study of TAP-144-SR (3M) to Evaluate Hormone Dynamics, Pharmacokinetics, Safety and Efficacy of TAP-144-SR (6M) 22.5 mg Subcutaneous Injection for 48 Weeks in Prostate Cancer Patients Previously Treated With Hormonal Therapy
Brief Title: A Phase 3 Comparative Study of TAP-144-SR(6M) in Prostate Cancer Patients Previously Treated With Hormonal Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP-144-SR(6M)IP/CPH-002; U1111-1128-6861 (Registry Identifier: WHO); JapicCTI-121763 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP-144-SR(6M) (Experimental): TAP-144-SR(6M) 22.5 mg, injection, treatment interval 24 weeks for up to 48 weeks.
  Interventions: Drug: TAP-144-SR(6M)
- TAP-144-SR(3M) (Active Comparator): TAP-144-SR(3M) 11.25 mg, injection, treatment interval 12 weeks for up to 48 weeks.
  Interventions: Drug: TAP-144-SR(3M)

INTERVENTIONS:
Drug: TAP-144-SR(6M)
  Arms: TAP-144-SR(6M)
Drug: TAP-144-SR(3M)
  Arms: TAP-144-SR(3M)

SUMMARY:
The purpose of this study is to evaluate hormone dynamics, pharmacokinetics, safety, and efficacy of TAP-144-SR(6M) against TAP-144-SR(3M) in prostate cancer patients previously treated with hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has histopathologically confirmed prostate cancer in Japanese.
2. The participant has prostate cancer in the clinical stages of T1b-T4, N-any and M-any by TNM classification on clinical diagnosis at the time of diagnosis.
3. The participant has ECOG performance status of grades 0, 1, or 2 at screening.
4. The participant with PSA level which has not increased 25 % or greater and 2 ng/mL or more from the nadir at the measurement points 4 weeks or longer apart within the screening period of 12 weeks.
5. Patients who receive the marketed product for 3 months (LEUPLIN SR FOR INJECTION KIT 11.25) at screening
6. Patients who have received the marketed products, TAP-144-SR (1M) and TAP-144-SR (3M), for 24-96 weeks in total at the scheduled starting date of the study drug, but not including administration period treated as neoadjuvant therapy for prostatectomy and/or radiation therapy
7. Patients who have continued the nonsteroidal antiandrogen for longer than 12 weeks at the scheduled starting date of the study drug, if a nonsteroidal antiandrogen is concomitantly administered
8. The participant with a serum testosterone level at screening < 100ng/dL
9. The participant meets the following criteria of renal, bone-marrow and hepatic functions on the laboratory test results at screening:

（1） Renal function: serum creatinine level< 1.5 times the upper limit of normal (ULN) （2） Bone-marrow function: white blood count ≥ 3,500/ mm3, platelet count ≥ 100,000/L, hemoglobin ≥ 10.0g/dL （3） Hepatic function: AST(GOT), ALT(GPT), ALP and total bilirubin ≤ 2.5 times the ULN 10. The participant's life expectancy is at least 24 months at informed consent.

Exclusion Criteria:

1. The participant has active multiple primary cancers, (synchronous multiple primary cancer or metachronous multiple primary cancer with the disease-free survival ≤ 5 years)
2. The participant has received surgical castration.
3. The participant has ever received LHRH agonists other than commercially available 1-month or 3-month depot of leuprolide acetate.
4. The participant has ever received LHRH antagonists.
5. Patients who have previously received estrogen preparations or corticosteroids for prostate cancer
6. Patients who have previously received chemotherapy for prostate cancer
7. Patients who are receiving or received the marketed product for 3 months (LEUPLIN SR FOR INJECTION KIT 11.25) or the marketed products for 1 month (LEUPLIN FOR INJECTION 3.75 and KIT 3.75) as an adjuvant therapy after prostatectomy and/or radiotherapy
8. Patients who are receiving or received the marketed product for 3 months (LEUPLIN SR FOR INJECTION KIT 11.25) for intermittent androgen deprivation therapy
9. Patients who received the following drugs within 24 weeks (168 days) after starting the study drug: Steroidal antiandrogens, type II 5α-reductase inhibitors
10. The participant received any of the following within 16 weeks (112 days) prior to study enrollment:

（1） Radiotherapy. As for I-125 brachytherapy, within 35 weeks (245 days) prior to study enrollment.

（2） Prostatectomy （3） Experimental therapy including high-intensity focused ultrasound therapy (HIFU), immunotherapy, and gene therapy 11. Patients who received the following drugs within 4 weeks (28 days) before starting the study drug: Testosterones, ketoconazole（except for external preparations）, spironolactone, corticosteroids (excluding their inhalants and external preparations), and Chinese medicines and dietary supplements containing saw palmetto 12. Patients whose QTcF interval exceeded 460 msec on the 12-lead electrocardiogram at screening 13. The participant has a history of hypersensitivity to synthetic LHRH, LHRH derivative or any component of the study drug.

14. The participant has central nervous system metastasis which requires treatment or which is symptomatic.

15. The participant already has a history or has a complication or may have renal disorder caused by spinal cord compression or ureteric obstruction.

16. The participant has a history of serious drug allergic reaction/hypersensitivity 17. The participant has a history of, or has been diagnosed with thromboembolism including myocardial infarction, cerebral infarction, venous thrombosis, and pulmonary embolism, or cardiac failure

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (16):
- Japan (16):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Fukuoka, Fukuoka
  - Maebashi, Gunma
  - Sapporo, Hokkaido
  - Kanazawa, Ishikawa-ken
  - Yokohama, Kanagawa
  - Sendai, Miyagi
  - Nigata-shi, Niigata
  - Osaka, Osaka
  - Suita-shi, Osaka
  - Ageo-shi, Saitama
  - Kita-adachi-gun, Saitama
  - Shizuoka, Shizuoka
  - Itabashi-ku, Tokyo
  - Shinjuku-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in Japan from 11 April 2012 to 04 April 2014.
Pre-assignment Details: Prostate cancer patients previously treated with hormonal therapy were enrolled in 1 of 2 treatment groups. Two patients withdrew from the period between randomization and starting study drugs (1 in TAP-144-SR(6M) arm and 1 in TAP-144-SR(3M) arm).
Period: Overall Study
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Started | 82 | 80
Received Study Drug | 81 | 79
Completed | 76 | 74
Not Completed | 6 | 6
Not completed — Adverse Event | 2 | 3
Not completed — Major Protocol Deviation | 1 | 1
Not completed — High Prostate specific antigen | 2 | 1
Not completed — Did Not Receive Study Drug | 1 | 1

BASELINE CHARACTERISTICS:
Population: The population included all participants who were randomized to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M) | Total
Number analyzed (Participants) | 82 | 80 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.3 (6.32) | 72.6 (6.49) | 73.0 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 82 | 80 | 162
Weight [Mean (Standard Deviation); unit: kg] | 64.03 (8.689) | 65.83 (8.098) | 64.92 (8.424)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.61 (2.731) | 24.32 (2.769) | 23.96 (2.764)
Gleason Score [Number; unit: Participants] — Gleason score is a score used in prostate cancer grading. Prostate cancer staging is the process by which physicians categorize the risk of cancer having spread beyond the prostate, or equivalently, the probability of being cured with local therapies such as surgery or radiation. Gleason score are often grouped into four stages (I-IV) of prostate cancer. Gleason scores range from 2 to 10, with 2 representing the most well-differentiated tumors and 10 the least-differentiated tumors.
  Participants
    2 | 0 (0.0) | 0 (0.0) | 0
    3 | 0 (0.0) | 0 (0.0) | 0
    4 | 0 (0.0) | 0 (0.0) | 0
    5 | 2 (2.4) | 2 (2.5) | 4
    6 | 8 (9.8) | 7 (8.8) | 15
    7 | 35 (42.7) | 29 (36.3) | 64
    8 | 14 (17.1) | 21 (26.3) | 35
    9 | 20 (24.4) | 21 (26.3) | 41
    10 | 3 (3.7) | 0 | 3
Tumor-node-metastasis (TNM) classification at diagnosis: T [Number; unit: Participants] — Number of participants for whom TNM classification at diagnosis: T data is available in the TAP-144-SR(3M) treatment arm is 79, respectively.
  The categories of T is ranged from T1 (better) to T4 (worse). Tx represents "tumor cannot be evaluated" and T0 represents "no signs of tumor."
  Participants
    T0 | 0 (0.0) | 0 (0.0) | 0
    T1 | 17 (20.7) | 16 (20.3) | 33
    T2 | 32 (39.0) | 24 (30.4) | 56
    T3 | 29 (35.4) | 33 (41.8) | 62
    T4 | 4 (4.9) | 6 (7.6) | 10
    TX | 0 (0.0) | 0 (0.0) | 0
    Unknown | 0 (0) | 0 (0.0) | 0
TNM classification at diagnosis: N [Number; unit: Participant] — Number of participants for whom TNM classification at diagnosis: N data is available in the TAP-144-SR(3M) treatment arm is 79, respectively. The categories of N is represented by Nx (lymph nodes cannot be evaluated), N0 (tumor cells absent from regional lymph nodes), and N1 (regional lymph node metastasis present).
  Participant
    N0 | 69 | 62 | 131
    N1 | 13 | 17 | 30
    NX | 0 | 0 | 0
    Unknown | 0 | 0 | 0
TNM classification at diagnosis: M [Number; unit: participants] — Number of participants for whom TNM classification at diagnosis: M data is available in the TAP-144-SR(3M) treatment arm is 79, respectively. The categories of M is represented by M0 (no distant metastasis), and M1 (metastasis to distant organs (beyond regional lymph nodes).
  participants
    M0 | 63 | 62 | 125
    M1 | 19 | 17 | 36
    Unknown | 0 | 0 | 0
Period between date of first dianosis and date of informed consent [Mean (Standard Deviation); unit: Years] | 1.653 (2.0866) | 1.748 (2.0410) | 1.700 (2.0583)
Period between first dose dates of leuproride acetate (over-the-counter) and the study drug [Mean (Standard Deviation); unit: Weeks] | 46.328 (20.0833) | 46.595 (20.8584) | 46.460 (20.4056)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — Number of participants for whom ECOG Performance Status data is available in Baseline Characteristics is 81 and 79 in each treatment arm, respectively. The categories of ECOG Performance Status is represented from 0 (Fully active, better) to 4 (Completely disabled, worse).
  Participants
    0 | 73 | 71 | 144
    1 | 7 | 7 | 14
    2 | 1 | 1 | 2
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Suppression of Serum Testosterone to Castrate Level
Description: Comparison of the proportion of patients maintained at castration level (≤100 ng/dL)
Time Frame: From the start of study drug administration through Week 48
Population: Full analysis set participants (all randomized participants who received at least 1 dose of study drug) was used.
Measure: Number; unit: Participants
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 81 | 79
Participants
  Number of participants maintained | 81 | 78
  Number of participants who did not maintain | 0 | 1

2. Secondary Outcome: Time Course of Changes in Serum Testosterone
Time Frame: From baseline to Week 48
Population: Full analysis set participants (all randomized participants who received at least 1 dose of open-label study drug) with both Baseline and a post-baseline value; last observation carried forward was used.
Measure: Median (Full Range); unit: ng/dL
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 81 | 79
ng/dL
  Baseline | 8.0 [0 to 33] | 7.0 [0 to 388]
  Week 1 | 6.0 [0 to 33] | 7.0 [0 to 267]
  Week 2 | 7.0 [0 to 37] | 6.0 [0 to 55]
  Week 4 | 7.0 [0 to 35] | 8.0 [0 to 33]
  Week 8 | 7.5 [0 to 53] | 8.0 [0 to 33]
  Week 12 | 7.0 [0 to 41] | 8.0 [0 to 36]
  Week 16 | 7.0 [0 to 45] | 7.5 [0 to 34]
  Week 20 | 8.0 [0 to 43] | 6.0 [0 to 40]
  Week 24 | 7.0 [0 to 37] | 6.0 [0 to 33]
  Week 25 | 6.0 [0 to 30] | 5.5 [0 to 30]
  Week 26 | 5.0 [0 to 35] | 4.0 [0 to 32]
  Week 28 | 8.0 [0 to 36] | 6.0 [0 to 36]
  Week 32 | 9.0 [0 to 41] | 8.0 [0 to 30]
  Week 36 | 8.0 [0 to 34] | 7.0 [0 to 40]
  Week 40 | 8.0 [0 to 39] | 8.0 [0 to 37]
  Week 44 | 7.0 [0 to 37] | 8.0 [0 to 33]
  Week 48 | 9.0 [0 to 42] | 6.0 [0 to 34]

3. Secondary Outcome: Time Course of Changes in Serum Luteinizing Hormone (LH)
Time Frame: From baseline to Week 48
Population: as for outcome 2
Measure: Median (Full Range); unit: mIU/mL
Units Other Than Participants: participants
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 81 | 79
mIU/mL
  Baseline | 0.000 [0.00 to 1.44] | 0.000 [0.00 to 12.25]
  Week 1 | 0.160 [0.00 to 1.03] | 0.220 [0.00 to 7.57]
  Week 2 | 0.180 [0.00 to 0.68] | 0.150 [0.00 to 2.91]
  Week 4 | 0.120 [0.00 to 0.37] | 0.110 [0.00 to 0.65]
  Week 8 | 0.000 [0.00 to 0.33] | 0.000 [0.00 to 0.67]
  Week 12 | 0.000 [0.00 to 0.35] | 0.110 [0.00 to 1.56]
  Week 16 | 0.000 [0.00 to 0.38] | 0.055 [0.00 to 0.87]
  Week 20 | 0.000 [0.00 to 0.36] | 0.110 [0.00 to 0.58]
  Week 24 | 0.000 [0.00 to 1.38] | 0.000 [0.00 to 0.63]
  Week 25 | 0.150 [0.00 to 0.67] | 0.185 [0.00 to 0.54]
  Week 26 | 0.170 [0.00 to 0.84] | 0.130 [0.00 to 0.48]
  Week 28 | 0.110 [0.00 to 0.35] | 0.000 [0.00 to 0.59]
  Week 32 | 0.000 [0.00 to 0.26] | 0.000 [0.00 to 0.66]
  Week 36 | 0.000 [0.00 to 0.24] | 0.000 [0.00 to 0.76]
  Week 40 | 0.000 [0.00 to 0.31] | 0.000 [0.00 to 0.49]
  Week 44 | 0.000 [0.00 to 0.32] | 0.000 [0.00 to 0.66]
  Week 48 | 0.000 [0.00 to 0.42] | 0.000 [0.00 to 0.84]

4. Secondary Outcome: Time Course of Changes in Serum Follicle-stimulating Hormone (FSH)
Time Frame: From baseline to Week 48
Population: as for outcome 2
Measure: Median (Full Range); unit: mIU/mL
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 81 | 79
mIU/mL
  Baseline | 5.120 [1.93 to 13.31] | 4.780 [2.02 to 18.52]
  Week 1 | 5.430 [1.87 to 15.52] | 4.810 [1.77 to 17.62]
  Week 2 | 4.890 [1.99 to 13.12] | 4.710 [1.81 to 16.40]
  Week 4 | 4.625 [1.72 to 14.11] | 4.950 [1.49 to 16.19]
  Week 8 | 5.225 [1.90 to 13.75] | 5.240 [1.79 to 17.23]
  Week 12 | 5.340 [2.24 to 14.04] | 5.110 [1.86 to 15.97]
  Week 16 | 5.300 [2.07 to 13.87] | 5.370 [1.81 to 15.65]
  Week 20 | 5.030 [1.65 to 12.21] | 5.260 [1.91 to 15.01]
  Week 24 | 4.990 [1.97 to 13.45] | 5.150 [2.12 to 16.47]
  Week 25 | 5.210 [2.16 to 12.92] | 4.970 [1.84 to 17.02]
  Week 26 | 5.010 [2.34 to 13.14] | 5.020 [1.96 to 14.69]
  Week 28 | 5.060 [2.31 to 13.38] | 5.070 [2.05 to 13.63]
  Week 32 | 5.210 [2.32 to 13.20] | 5.030 [2.08 to 12.54]
  Week 36 | 5.585 [2.01 to 13.00] | 4.970 [2.09 to 14.08]
  Week 40 | 5.100 [1.80 to 14.85] | 4.910 [2.05 to 13.20]
  Week 44 | 5.150 [1.69 to 12.90] | 4.990 [2.17 to 14.14]
  Week 48 | 5.110 [1.44 to 11.69] | 4.820 [2.18 to 14.46]

5. Secondary Outcome: Time Course of Change Rate in Serum PSA (FAS)
Description: Evaluation according to the "Criteria for therapeutic effect" from the General Rule for Clinical Pathological Studies on Prostate Cancer, 4th edition (determination of therapeutic effect by prostate-specific antigen [PSA])
Time Frame: From baseline to Week 48
Population: as for outcome 2
Measure: Median (Full Range); unit: percent change
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 81 | 79
percent change
  Week 4 | -7.930 [-100.00 to 181.82] | -10.000 [-100.00 to 122.95]
  Week 8 | -14.255 [-100.00 to 190.06] | -15.880 [-100.00 to 184.85]
  Week 12 | -20.810 [-100.00 to 360.84] | -21.130 [-100.00 to 754.55]
  Week 16 | -19.720 [-100.00 to 634.69] | -20.650 [-100.00 to 1866.67]
  Week 20 | -44.740 [-100.00 to 932.65] | -39.970 [-100.00 to 3718.18]
  Week 24 | -49.270 [-100.00 to 2002.04] | -31.110 [-100.00 to 9900.00]
  Week 28 | -56.705 [-100.00 to 2920.41] | -45.875 [-100.00 to 15354.55]
  Week 32 | -57.690 [-100.00 to 7389.80] | -40.745 [-100.00 to 21051.52]
  Week 36 | -60.710 [-100.00 to 9675.51] | -50.520 [-100.00 to 23506.06]
  Week 40 | -80.610 [-100.00 to 5348.98] | -58.520 [-100.00 to 21627.27]
  Week44 | -74.105 [-100.00 to 6859.18] | -54.585 [-100.00 to 24506.06]
  Week 48 | -72.900 [-100.00 to 6818.37] | -59.400 [-100.00 to 22839.39]

6. Secondary Outcome: The Maximum Rate of Change in PSA Suppression (FAS)
Description: Evaluation according to the "Criteria for therapeutic effect" from the General Rule for Clinical Pathological Studies on Prostate Cancer, 4th edition (determination of therapeutic effect by PSA)
Time Frame: From baseline to Week 48
Population: as for outcome 2
Measure: Median (Full Range); unit: percent change
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 54 | 55
percent change | -86.225 [-100.00 to 108.73] | -67.030 [-100.00 to 75.76]

7. Secondary Outcome: Percentage of Participants With Progression by PSA (FAS)
Description: as for outcome 6
Time Frame: From baseline to Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Units Other Than Participants: Participants
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 80 | 77
percentage of participants
  Presence of disesase progression: Yes | 7.5 | 92.5
  Presence of disesase progression: No | 6.5 | 93.5

8. Secondary Outcome: Soft Tissue Response
Description: Assessment in accordance with the "criteria for therapeutic effect" from the General Rule for Clinical Pathological Studies on Prostate Cancer, 4th edition. Soft tissue response was evaluated in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: At week 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 79 | 76
Percentage of participants
  Complete response | 0.0 | 0.0
  Partial Response | 0.0 | 0.0
  Stable Disease | 13.9 | 11.8
  Progressive Disease | 0.0 | 2.6
  Not Evaluable | 86.1 | 85.5

9. Secondary Outcome: Bone Lesion Response
Description: Partially revised assessment based on the "criteria for therapeutic effect" from the General Rule for Clinical and Pathological Studies on Prostate Canter, 4th edition. Response is measured using bone scintigraphy. Increase in new (2 or more) bone lesion is considered as progression
Time Frame: At Week 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 78 | 75
Percentage of participants
  Presence of disesase progression: New lesions ≥ 2 | 1.3 | 1.3
  Presence of disesase progression: New lesions < 1 | 98.7 | 98.7

10. Secondary Outcome: Serum Unchanged TAP-144 Level
Time Frame: From baseline to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 81 | 79
ng/dL
  Baseline | 0.07113 (0.043808) | 0.06188 (0.035339)
  Week 1 | 0.1304 (0.16388) | 0.1869 (0.077198)
  Week 2 | 0.3085 (0.30523) | 0.1335 (0.083060)
  Week 4 | 0.8845 (0.52695) | 0.1132 (0.12110)
  Week 8 | 0.1792 (0.10354) | 0.08374 (0.041078)
  Week 12 | 0.1256 (0.068860) | 0.08039 (0.056305)
  Week 16 | 0.1024 (0.093951) | 0.1220 (0.067137)
  Week 20 | 0.06957 (0.053682) | 0.08450 (0.039532)
  Week 24 | 0.05167 (0.043221) | 0.07437 (0.045186)
  Week 25 | 0.1353 (0.29809) | 0.1978 (0.083286)
  Week 26 | 0.4318 (0.63101) | 0.1418 (0.087312)
  Week 28 | 0.7622 (0.42483) | 0.1067 (0.054505)
  Week 32 | 0.1524 (0.098308) | 0.08236 (0.046180)
  Week 36 | 0.1091 (0.057582) | 0.08407 (0.075147)
  Week 40 | 0.09118 (0.065771) | 0.1086 (0.051455)
  Week 44 | 0.06958 (0.055624) | 0.08639 (0.051923)
  Week 48 | 0.04596 (0.030006) | 0.07945 (0.066980)

11. Secondary Outcome: 12-lead ECG
Time Frame: At 1 hour, week 24, and week 48 after administration
Population: Safety evaluation was conducted in the safety analysis set (SAS), which includes all 160 patients who received the study drug [TAP-144-SR (&M) group: 81 patients, TAP-144-SR (3M) group: 79 patients
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Number analyzed (Participants) | 81 | 79
msec
  QTcF interval measurement at Basline | 429.0 (15.75) | 436.2 (15.63)
  QTcF interval measurement at 1 hour | 422.2 (20.80) | 432.2 (21.93)
  QTcF interval measurement at Week 24 | 425.0 (20.01) | 433.4 (18.91)
  QTcF interval measurement at Week 48 | 428.1 (16.42) | 431.7 (16.05)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 14 days (or 30 days for a serious adverse event) after the last dose of open-label study drug (up to 56 weeks).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAP-144-SR(6M) | TAP-144-SR(3M)
Serious Adverse Events (participants affected / at risk) | 10/81 | 8/79
Other Adverse Events (participants affected / at risk) | 74/81 | 71/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAP-144-SR(6M) (N=81) | TAP-144-SR(3M) (N=79)
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Dementia with Lewy bodies (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Disuse syndrome (General disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAP-144-SR(6M) (N=81) | TAP-144-SR(3M) (N=79)
Injection site induration (General disorders) | 14 | 11
Constipation (Gastrointestinal disorders) | 3 | 5
Dental caries (Gastrointestinal disorders) | 6 | 1
Injection site erythema (General disorders) | 12 | 6
Injection site pain (General disorders) | 6 | 5
Nasopharyngitis (Infections and infestations) | 18 | 25
Fall (Injury, poisoning and procedural complications) | 6 | 3
Contusion (Injury, poisoning and procedural complications) | 6 | 1
Blood creatine phosphokinase increased (Investigations) | 5 | 7
Weight increased (Investigations) | 1 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 3 | 5
Hot flush (Vascular disorders) | 5 | 5
Hypertension (Vascular disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.